CLINICAL TRIAL: NCT04027712
Title: High On-treatment Platelet Reactivity, Increased B-amyloid and Downregulation of MOTS-c Predict Mortality in Patients With Coronary Artery Disease and Type 2 Diabetes Mellitus: a 2-year Follow up Study
Brief Title: Platelet Reactivity, B-amyloid, MOTS-c and Mortality of Type II Diabetics With CAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Ignatios Ikonomidis,MD,PhD,FESC, Associate Professor of Cardiology, Director of Echocardiography and the Laboratory of Preventive Cardiology, 2nd Cardiology Department, National and Kapodistrian University of Athens, University of Athens
Other Study IDs: LTA_MOTS-c_bamyloid_DM_CAD
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Clopidogrel Resistance; Amyloid; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Alzheimer Disease; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fresh plasma, frozen plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Increased circulating b-amyloid and decreased Mitochondrial-derived peptide (MOTS-c), a peptide improving tissue insulin sensitivity, are reported in diabetes. The investigators plan to investigate the association of both biofactors with high on-clopidogrel platelet reactivity and cardiovascular mortality in type 2 diabetic patients with Coronary artery disease

DETAILED DESCRIPTION:
In type II diabetic patients with Coronary artery disease treated with clopidogrel and aspirin, the investigators plan to measure: i. maximum platelet aggregation to adenosine diphosphate (ADP) by Light Transmission Aggregometry (LTAmax), as a marker of on-clopidogrel treatment platelet reactivity ii. Malondialdehyde (MDA), as oxidative stress marker, Mitochondrial-derived peptide MOTS-c and b-amyloid. blood levels.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients with coronary artery disease, documented by coronary angiography,
* both per os or/and parenteral antidiabetic medications and double antiplatelet therapy (DAPT), constituted by a daily dose of 100 mg acetylsalicylic acid per os and a daily dose of 75 mg clopidogrel per os should be prescribed to the patients for at least one month before inclusion in the study

Exclusion Criteria:

* abnormal renal function (creatinine> 2.5 mg / dl),
* hepatic failure (bilirubin> 2 mg / dl),
* active malignancy,
* patients treated with drugs that affect platelet function, besides aspirin 100 mg qd and clopidogrel 75 mg qd,
* patients with a history of hemorrhagic mood,
* patients with thrombocytopenia (PLTs < 100x109 / L) and
* anemia (HCT <28%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetic patients with coronary artery disease, documented by coronary angiography, both per os or/and parenteric antidiabetic medications and double antiplatelet therapy (DAPT), constituted by a daily dose of 100 mg acetylsalicylic acid per os and a daily dose of 75 mg clopidogrel per os should be prescribed to the patients for at least one month before inclusion in the stud
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
mots-c predicts cardiovascular mortality in diabetic with coronary artery disease | 2 year follow up
  mots-c concentration in Diabetic with coronary artery disease treated with acetyl-salicylic and clopidogrel predicts cardiovascular mortality
b amyloid predicts cardiovascular mortality in diabetic with coronary artery disease | 2 year follow up
  b amyloid concentration in Diabetic with coronary artery disease treated with acetyl-salicylic and clopidogrel predicts cardiovascular mortality
b amyloid predicts cardiovascular mortality in diabetic with coronary artery | 2 year follow up
  Resistance to clopidogrel as defined by Light Transmission Aggregometry in diabetic with coronary artery disease treated with acetyl-salicylic and clopidogrel predicts cardiovascular mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, AssProfessor, Study Chair — University of Athens
Locations (1):
- General & University Hospital "Attikon", Chaïdári, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ikonomidis I, Katogiannis K, Kyriakou E, Taichert M, Katsimaglis G, Tsoumani M, Andreadou I, Maratou E, Lambadiari V, Kousathana F, Papadopoulou A, Varlamos C, Plotas P, Parissis J, Stamatelopoulos K, Alexopoulos D, Dimitriadis G, Tsantes AE. beta-Amyloid and mitochondrial-derived peptide-c are additive predictors of adverse outcome to high-on-treatment platelet reactivity in type 2 diabetics with revascularized coronary artery disease. J Thromb Thrombolysis. 2020 Apr;49(3):365-376. doi: 10.1007/s11239-020-02060-4. PMID 32052315